CLINICAL TRIAL: NCT02648464
Title: Hydroxychloroquine for the Prevention of Recurrent Cardiovascular Events in Myocardial Infarction Patients - a Safety Pilot Trial
Brief Title: Hydroxychloroquine for the Prevention of Cardiovascular Events in Myocardial Infarction Patients - a Safety Pilot Trial
Acronym: OXI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Finnish Foundation for Cardiovascular Research (Other); Orion Corporation, Orion Pharma (Industry); Aarne Koskelo Foundation (Other); Finnish Cultural Foundation (Other)
Responsible Party: Principal Investigator, Otto Hartman, MD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015-000233-73
Record Dates: First submitted 2015-12-18; First posted 2016-01-07 (Estimated); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Myocardial Infarction; Acute Coronary Syndrome; Inflammation; Hydroxychloroquine; Antirheumatic Agents; Cardiovascular Diseases
Keywords: Hydroxychloroquine; anti-inflammatory; Myocardial infarction; cardiovascular diseases
MeSH Terms: conditions — Myocardial Infarction; Acute Coronary Syndrome; Inflammation; Cardiovascular Diseases | interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydroxychloroquine (Experimental): Hydroxychloroquine 300 mg tablet by mouth daily for 6 months. Patients under the weight of 60 kg: hydroxychloroquine 300 mg tablet daily for 5 days per week for 6 months.
  Interventions: Drug: Hydroxychloroquine
- Placebo (Placebo Comparator): Placebo tablet by mouth daily for 6 months. Patients under the weight of 60 kg: placebo tablet daily for 5 days per week for 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine
  Other Names: Oxiklorin
  Arms: Hydroxychloroquine
Drug: Placebo
  Arms: Placebo

SUMMARY:
This safety pilot study evaluates the effect of hydroxychloroquine on preventing recurrent cardiovascular events among myocardial infarction patients. Half of the participants will receive hydroxychloroquine, whereas the other half will receive placebo during six months.

DETAILED DESCRIPTION:
Anti-rheumatic medications decrease cardiovascular mortality in rheumatoid arthritis patients, based mainly on their anti-inflammatory effect. No studies have addressed their effect on preventing recurrent cardiovascular events among non-rheumatic patients.

In the pilot phase 200 myocardial infarction patients will be recruited during their index visit to the study hospitals. Patients will be randomized after initial coronary angiography to receive either hydroxychloroquine 300 mg a day or placebo during six months. Patients will be followed up until 12 months at four visits. Visit one is at doctor´s office at 3 to 5 weeks from the day of recruitment. Visit two is at study nurse´s office at 5.5 to 6 months. Visit three is a phone interview by the study nurse at 8.5 to 9.5 months. Visit four at 11.5 to 12.5 months is at doctor´s office.

This study evaluates the safety of hydroxychloroquine in the setting of myocardial infarction, and whether hydroxychloroquine treatment could reduce the incidence of recurrent cardiovascular events among myocardial infarction patients. Furthermore, the effect of hydroxychloroquine on cardiovascular risk factors and systemic inflammation parameters will be studied. In a subgroup of 40 patients, the effect of hydroxychloroquine on aortic inflammation will be assessed by PET/CT scan.

If this safety pilot study with 200 patients proves successful (i.e. no major complications), 2500 patients will be recruited in additional centers in Finland and the Nordic Countries.

Orion Pharma provides the active hydroxychloroquine tablet (Oxiklorin) but provides no other assistance or funding for the study.

ELIGIBILITY:
Inclusion Criteria:

Patients must have high-sensitivity troponin or CKMB above the upper limit of normal with at least one of the following criteria:

1. Anginal symptoms suggestive of cardiac ischemia

   1. Accelerating pattern of anginal pain (episodes of angina that have at least 5 minutes duration and are more frequent, severe, longer in duration and/or precipitated by less exertion).
   2. Prolonged (>20 minutes) or recurrent anginal pain at rest or with minimal effort.
   3. Anginal pain at rest or with minimal exertion, and at least 20 minutes of duration, occurring >48 hours after an acute Q-wave myocardial infarction.
2. ECG criteria

   1. New, persistent or transient ST-segment depression >0,1 mV (0,08 seconds after the J-point) in at least 2 extremity leads or 3 precordial leads.
   2. New, persistent or transient ST-segment elevation in two contiguous leads ≥0.2 mV in men or ≥0.15 mV in women in leads V2-V3, and/or ≥0.1 mV in other leads.

Patients will be enrolled within 96 hours of coronary angiography

Exclusion Criteria:

* Contraindication for hydroxychloroquine (porphyria, psoriasis, retinopathy, hypersensitivity)
* Rheumatoid arthritis or other rheumatic disease
* Significant neuropathy of any cause
* Cardiomyopathy (diagnosed before the onset of index hospitalization)
* Muscle disease (that could worsen by the use of hydroxychloroquine)
* Pregnant or nursing women, and women of childbearing potential without efficient contraceptives.
* Angina precipitated by obvious provoking factors
* Prolonged ECG's corrected QT interval (>480 ms)
* Ongoing antibiotic therapy of any duration
* Uncontrolled severe cardiac arrhythmia resulting in hemodynamic instability
* Severe hepatic failure (alanine transaminase or gamma-glutamyltransferase ≥2 times above normal limits or international normalized ratio (INR) >1,5 and patient not using warfarin, and due to other than cardiac reasons).
* Renal failure, glomerular filtration rate <50 ml/min/1,73m2
* Hemoglobin <100 g/l (if not possible to correct with transfusion)
* Planned percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG)
* Index myocardial infarction due to PCI or CABG restenosis.
* Inability to interpret ST-T segment changes on ECG (e.g. complete left bundle branch block or paced rhythm)
* Prior thrombolytic therapy (within 12 hours)
* Inability to give informed consent
* Fulminant vomiting or other disability to give oral medication
* Over 80 years of age
* Life expectancy less than one year
* Receiving another investigational drug within 4 weeks prior to the study. (Patients who have participated in investigational trials before the 4-week time period may be randomized as long as they have reached the primary endpoint).
* Patients with any other medical condition which, in the investigator's opinion, would interfere with optimal participation in the study or produce a significant risk to the patient

In addition, patients are not eligible for the PET/CT subgroup if they have received statin-therapy in the last 2 months prior to the hospitalization (i.e. statin therapy started during the index hospitalization is not an exclusion criteria).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of major cardiovascular adverse events | Twelve months
  Myocardial infarction, mortality, hospitalization for unstable angina, and heart failure

SECONDARY OUTCOMES:
Rate of the primary endpoint plus stroke and urgent coronary revascularization | Twelve months
Effect on the incidence of type 2 diabetes and the level of Hba1c | Six months
Effect on cholesterol levels | Six months
  The effect of hydroxychloroquine on total cholesterol, low-density lipoprotein, high-density lipoprotein, and triglyceride levels
Effect on high-sensitivity C-reactive protein (hs-CRP) level | Six months
Effect on soluble biomarkers of inflammation | Six months
  Frozen samples (plasma and whole blood) will be stored for future evaluation of biomarkers related to inflammation and cardiovascular disease, such as tumor necrosis factor alpha, interleukin 6 (IL-6), IL-1beta, IL-18, and messenger ribonucleic acid (mRNA) analyses.
Effect on aortic inflammation assessed by PET / CT scan | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Juha Sinisalo, Professor, Study Director — Helsinki University Central Hospital
Locations (6):
- Finland (6):
  - Helsinki University Central Hospital, Helsinki
  - North Karelia Central Hospital, Joensuu
  - Kymenlaakso Central Hospital, Kotka
  - Päijät-Häme Central Hospital, Lahti
  - South Karelia Central Hospital, Lappeenranta
  - South Ostrobotnia Central Hospital, Seinäjoki

IPD SHARING:
Plan to Share IPD: Yes
Study data is planned to be available at the study organization´s website, and by specific request from the investigator

REFERENCES:
- [Background] Hartman O, Kovanen PT, Lehtonen J, Eklund KK, Sinisalo J. Hydroxychloroquine for the prevention of recurrent cardiovascular events in myocardial infarction patients: rationale and design of the OXI trial. Eur Heart J Cardiovasc Pharmacother. 2017 Apr 1;3(2):92-97. doi: 10.1093/ehjcvp/pvw035. PMID 28025216
- [Derived] Simonen P, Ulander L, Eklund KK, Niemi M, Backman JT, Gylling H, Sinisalo J; OXI pilot trial. The effect of hydroxychloroquine on cholesterol synthesis depends on the profile of cholesterol metabolism. A controlled clinical study. Atheroscler Plus. 2024 Mar 1;55:93-97. doi: 10.1016/j.athplu.2024.02.002. eCollection 2024 Mar. PMID 38487037
- [Derived] Ulander L, Simonen P, Tolppanen H, Hartman O, Rissanen TT, Eklund KK, Kalaoja M, Kurkela M, Neuvonen M, Niemi M, Backman JT, Gylling H, Sinisalo J; OXI pilot trial. The effect of hydroxychloroquine on cholesterol metabolism in statin treated patients after myocardial infarction. Atheroscler Plus. 2023 Jun 26;53:26-32. doi: 10.1016/j.athplu.2023.06.003. eCollection 2023 Sep. PMID 37448694